CLINICAL TRIAL: NCT01464411
Title: Phase II Clinical Trial of Dasatinib First Line Therapy for Patients With Newly Diagnosed Chronic Myeloid Leukemia in Chronic Phase
Brief Title: Dasatinib in Newly Diagnosed Chronic-Phase Chronic Myeloid Leukemia in Japan
Acronym: D-First
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kanto CML Study Group (Other)
Responsible Party: Principal Investigator, Takashi Kumagai, M.D, Ph.D, Kanto CML Study Group
Other Study IDs: KCSG-03
Record Dates: First submitted 2011-09-18; First posted 2011-11-03 (Estimated); Last update posted 2011-11-03 (Estimated); Status verified 2011-11

CONDITIONS: Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelogenous Leukemia, Chronic, Chronic Phase
Keywords: chronic myelogenous leukemia; chronic phase; Phase II; dasatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Copy numbers of bcr-abl mRNA in patients with dasatinib treatment will be measured by real-time RT-PCR to evaluate the efficiency of dasatinib.
  For patients resistant to dasatinib therapy, DNA mutation analysis of the bcr-abl gene associated with drug-resistancy will be performed.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate effectiveness of Dasatinib as the first line therapy for patients with newly diagnosed chronic myeloid leukemia in chronic phase in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed Chronic Myeloid Leukemia in the Chronic Phase
* 20 years old over
* ECOG performance status (PS) score 0-2
* Adequate organ function (hepatic, renal and lung)
* Signed written informed consent

Exclusion Criteria:

* A case with the double cancer of the activity
* Women who are pregnant or breastfeeding
* The case of Pleural effusion clearly
* Patients with complications or a history of severe or uncontrolled cardiovascular failure following

  * have a Myocardial infarction whithin 6 months
  * have an Angina within 3 months
  * have a Congestive heart failure within 3 months
  * have a QTc interval of more than 450msec at baseline
* A serious uncontrolled medical disorder that would impair the ability of the subjects to receive protocol therapy

Min Age: 20 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed chronic-phase chronic myelogenous leukemia in Japan
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2011-07

PRIMARY OUTCOMES:
Rate of complete molecular response (CMR) after treatment with dasatinib | by 18 months
  The rate(%) of patients who achieve complete molecular response (CMR) by 18 months after the dasatinib therapy will be measured to evaluate the efficiency of dasatinib.

SECONDARY OUTCOMES:
complete molecular response (CMR) | by 3,6,12,24, 36 months
Major Molecular Response(MMR) | by 3,6,12,18,24,36 months
Complete Cytogenetic Response(CCyR) | by 6,12 months
Expansions rate of large granular lymphocyte | by 12 months
Progression free survival | at 36 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | by 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kanto CML Study Group, Tokyo, Japan

REFERENCES:
- [Derived] Iriyama N, Fujisawa S, Yoshida C, Wakita H, Chiba S, Okamoto S, Kawakami K, Takezako N, Kumagai T, Inokuchi K, Ohyashiki K, Taguchi J, Yano S, Igarashi T, Kouzai Y, Morita S, Sakamoto J, Sakamaki H. Early cytotoxic lymphocyte expansion contributes to a deep molecular response to dasatinib in patients with newly diagnosed chronic myeloid leukemia in the chronic phase: results of the D-first study. Am J Hematol. 2015 Sep;90(9):819-24. doi: 10.1002/ajh.24096. PMID 26103598
- [Derived] Iriyama N, Fujisawa S, Yoshida C, Wakita H, Chiba S, Okamoto S, Kawakami K, Takezako N, Kumagai T, Inokuchi K, Ohyashiki K, Taguchi J, Yano S, Igarashi T, Kouzai Y, Morita S, Sakamoto J, Sakamaki H. Shorter halving time of BCR-ABL1 transcripts is a novel predictor for achievement of molecular responses in newly diagnosed chronic-phase chronic myeloid leukemia treated with dasatinib: Results of the D-first study of Kanto CML study group. Am J Hematol. 2015 Apr;90(4):282-7. doi: 10.1002/ajh.23923. Epub 2015 Mar 2. PMID 25530131